CLINICAL TRIAL: NCT05218642
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 2 Study in Male Subjects With Androgenetic Alopecia to Evaluate the Efficacy, Safety, and Tolerability of KX-826 Following Topical Multiple Dose Administration
Brief Title: To Evaluate Efficacy, Safety, and Tolerability of KX-826 in Male Subjects With Androgenetic Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KX0826-US-1003
Record Dates: First submitted 2022-01-30; First posted 2022-02-01 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-06

CONDITIONS: Alopecia; Male Pattern Hair Loss
Keywords: Androgenetic Alopecia; Hair loss; Hair thinning; Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): KX-826: 2.5mg twice daily
  Interventions: Drug: KX- 826 dosed at 2.5mg
- Arm B (Experimental): KX-826: 5mg once daily
  Interventions: Drug: KX-826 dosed at 5mg
- Arm C (Experimental): KX-826: 5mg twice daily
  Interventions: Drug: KX-826 dosed at 5mg
- Arm D (Experimental): Matching placebo to KX-826
  Interventions: Drug: Matching placebo to KX-826

INTERVENTIONS:
Drug: KX- 826 dosed at 2.5mg — 2.5mg of the investigational drug to be applied topically to scalp twice daily for 24 weeks
  Arms: Arm A
Drug: KX-826 dosed at 5mg — 5mg of the investigational drug to be applied topically to scalp once daily for 24 weeks
  Arms: Arm B
Drug: KX-826 dosed at 5mg — 5mg of the investigational drug to be applied topically to scalp twice daily for 24 weeks
  Arms: Arm C
Drug: Matching placebo to KX-826 — Placebo applied topically to scalp twice daily or once daily for 24 weeks
  Arms: Arm D

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, parallel group, phase 2 study to evaluate the efficacy, safety and tolerability of KX-826 in male subjects with androgenetic alopecia.

DETAILED DESCRIPTION:
KX-826 is a new investigational androgen receptor (AR) antagonist for the treatment of male pattern hair loss (androgenetic alopecia). A total of 120 subjects will be randomized to one of four cohorts: 2.5 mg BID, 5 mg QD, 5mg BID of KX-826 or placebo (BID or QD) for 24 weeks. The primary endpoint of the study is to assess the changes from baseline in non-vellus TAHC （Target Area Hair Counts）at Week 24 in comparison to placebo

ELIGIBILITY:
Inclusion Criteria:

1. Subject is capable of giving informed consent and complying with study procedures;
2. Subject is male between the ages of 18 and 70 years, inclusive;
3. Subject has a clinical diagnosis of mild to moderate androgenetic alopecia; rating IIIv, IV and V on the Norwood Hamilton Scale, with a history of ongoing hair loss;
4. Subject is willing to maintain the same hairstyle, hair length, and hair color throughout the study
5. Subject agrees to continue his other general hair care products and regimen for the entire study;
6. Subject is considered healthy by the Principal Investigator, based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG and vital signs (systolic blood pressure ≥90 and

   ≤150 mmHg, diastolic blood pressure ≥50 and ≤95 mmHg and pulse rate

   ≥45 and ≤100 bpm; one repeat of results is allowed to evaluate out of range values);
7. Negative COVID-19 results within 3 days prior first dosing

Exclusion Criteria:

1. Subject has any dermatological disorders of the scalp in the target region with the possibility of interfering with the application of the investigational drug, such as fungal or bacterial infections, seborrheic dermatitis, psoriasis, eczema, folliculitis, scars, or scalp atrophy;
2. Subject has any skin pathology or condition that, in the investigator's opinion, could interfere with the evaluation of the investigational drug or requires use of interfering topical, systemic (e.g., uncontrolled thyroid disease, certain genetic disorders that involve hair growth or patterns), or surgical therapy;
3. Subject has current or recent history (within 12 months) of hair weaves, non-breathable wigs, or hair bonding;
4. Subject had scalp hair transplants at any time
5. Subject has a history or active hair loss due to diffuse telogen effluvium, alopecia areata, scarring alopecia, trichotillomania, or conditions/ diseases other than AGA;
6. Subject has a current or recent history (within six months) of severe dietary or weight changes or has a history of eating disorder(s); if such has resulted in hair loss;
7. Any disorder, including but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

   * Affect the safety of the subject throughout the study
   * Influence the findings of the studies or their interpretations
   * Impede the subject's ability to complete the entire duration of study
8. Subject is currently enrolled in an investigational drug or device study;
9. Subject has used an investigational drug or investigational device treatment within 30 days prior to randomization;
10. Subject is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function;
11. Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse (defined as any illicit drug use), or subjects who are unable to return for scheduled follow-up visits;
12. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody;
13. Subject has a known hypersensitivity or previous allergic reaction to any of the active or inactive ingredients in the investigational drug or tattoo ink.
14. Subject has used any of the following topical preparations or procedures on the scalp:

    * Topical scalp treatments for hair growth including minoxidil, hormone therapy, anti-androgens, or other agents that are known to affect hair growth within 12 weeks of randomization;
    * Use of hair regrowth products, including minoxidil, for >4 continuous weeks within 6 months before randomization;
    * Medical shampoos or solutions which include Ketoconazole or the like (e.g. Terzolin) within four weeks prior to randomization;
    * Topical scalp over-the-counter (OTC) or cosmetic treatments known or reasonably believed to affect hair growth (e.g., brands such as Aminexil, Maxilene, Nioxin, Foltene, etc.) or hair health or hair growth products with saw palmetto, copper, etc. within four weeks of randomization;
    * Topical scalp treatments that may have ancillary effect on hair growth including, but not limited to, corticosteroids, pimecrolimus, tacrolimus, and retinoids within four weeks of randomization;
    * Scalp procedures (surgical, laser, light, or energy treatments, microneedling, etc.) within six months of randomization;
    * Platelet rich plasma (PRP) procedure on the scalp at any time point.
15. Subject has used the following systemic medications or procedures:

    * Beta blockers, cimetidine, diazoxide, or corticosteroids (including intramuscular and intralesional injections) within 12 weeks of randomization. Inhaled, intranasal, or ocular corticosteroids are allowed if use is stable [defined as doses and frequency unchanged for at least four weeks prior to randomization];
    * Retinoid, isotretinoin, vitamin A intake above 10,000 IU per day, or cyclosporine therapy within six months of randomization;
    * Use of immunoglobulins/immunomodulators (eg, cyclosporin) for >4 continuous weeks within 6 months of randomization,
    * Use of 5-α-reductase inhibitors (eg, finasteride or dutasteride) and/ or antiandrogens within 12 months before randomization;
    * Use of systemic cimetidine or ketoconazole for >2 continuous weeks within 3 months before randomization;
    * Chemotherapy or cytotoxic agents within 12 months of randomization;
    * Radiation of the scalp at any time point;
    * Use of systemic corticosteroids within 2 months of randomization for >2 consecutive weeks,
    * Other systemic therapy, which in the opinion of the investigator, may materially affect the subject's hair or hair growth, including, but not limited to, vitamin or homeopathy supplement hair growth or hair health products or other steroid hormones (in any form), including anabolic steroids;
16. An unwillingness of male participants to use highly effective contraceptive measures if engaging in sexual intercourse with a female partner of childbearing potential. Highly effective measures include use of a condom and spermicide and, for female partners, use of an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, progesterone subdermal implants, or a tubal ligation.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Assessment of change in Target Area Hair Counts | 24 weeks
  Changes from baseline in non-vellus TAHC (Target Area Hair Counts) in comparison to placebo

SECONDARY OUTCOMES:
Assessment of change in Hair Growth Assessment score | 6,12,18 and 24 weeks
  Changes from baseline in HGA (Hair Growth Assessment) score by Principal Investigator, subjects, and Canfield Independent panel review in comparison to placebo

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - First OC Dermatology, Fountain Valley, California
  - Qway Research LLC, Hialeah, Florida
  - Evoution Clinical Trials, Hialeah Gardens, Florida
  - Anchor Medical Research, LLC, Miami, Florida
  - Innovation Medical Group, LLC, Palmetto Bay, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - DelRicht Research, Baton Rouge, Louisiana
  - ALLCUTIS Research, LLC, Beverly, Massachusetts
  - ALLCUTIS Research, LLC, Portsmouth, New Hampshire
  - Clinical Trials of Texas, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided